CLINICAL TRIAL: NCT00059865
Title: Phase I/II Trial Of Gemcitabine And ALIMTA In Patients With Measurable Or Evaluable, Unresectable Or Metastatic Biliary Tract Carcinoma (Intrahepatic, Extrahepatic, Ampulla Or Vater) And Gallbladder Carcinoma
Brief Title: Gemcitabine Plus Pemetrexed Disodium in Treating Patients With Unresectable or Metastatic Biliary Tract or Gallbladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N9943; NCCTG-N9943; CDR0000298862 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02530 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: advanced adult primary liver cancer; unresectable gallbladder cancer; unresectable extrahepatic bile duct cancer; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed + gemcitabine (Experimental): Phase II: Patients receive pemetrexed disodium as in phase I and gemcitabine at the recommended phase II dose.
  Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine work in different ways to stop tumor cells from dividing so they stop growing or die. Pemetrexed disodium may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining gemcitabine with pemetrexed disodium may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gemcitabine when given together with pemetrexed disodium to see how well it works in treating patients with unresectable or metastatic biliary tract or gallbladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gemcitabine when administered with pemetrexed disodium in patients with unresectable or metastatic biliary tract or gallbladder cancer. (Phase I closed to accrual as of Oct. 2005.)
* Determine the 6-month survival rate of patients treated with this regimen.
* Determine the best objective tumor response rate and duration of best objective tumor response in patients treated with this regimen.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the individual patient variation in toxicity of and/or response to this regimen due to genetic differences in proteins involved in drug response in these patients.

OUTLINE: This is a multicenter phase I dose-escalation study of gemcitabine followed by a phase II study.

* Phase I: Patients receive pemetrexed disodium IV over 10 minutes and gemcitabine IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity (phase I closed to accrual as of October 2005).

Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive pemetrexed disodium as in phase I and gemcitabine at the recommended phase II dose.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 85 patients will be accrued for this study.

ELIGIBILITY:
* One of the following histologically or cytologically confirmed cancers not amenable to treatment with combined chemotherapy and radiotherapy:

  * Biliary tract (intrahepatic, extrahepatic, or ampulla of Vater) carcinoma
  * Gallbladder carcinoma
* Unresectable or metastatic disease
* No CNS metastases

  * Prior brain metastases treated with surgery or radiosurgery allowed provided treatment was completed at least 4 weeks ago and there is no evidence of CNS progression
* No clinically significant pericardial or pleural effusion or ascites unless able to be drained before study entry
* Performance status - ECOG 0-2
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST no greater than 5 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* Able to tolerate folic acid, corticosteroids, or cyanocobalamin supplements
* More than 4 weeks since prior biologic or immunologic therapy
* No prior biologic or immunologic therapy for metastatic disease
* No concurrent immunotherapy
* No concurrent colony-stimulating factors during course 1
* No prior chemotherapy for metastatic disease
* No prior gemcitabine
* Prior chemoembolization allowed provided the following are true:

  * At least 4 weeks since prior chemoembolization
  * Evidence of new tumor growth since therapy
* At least 6 months since prior chemotherapy used as a radiosensitizer (in adjuvant setting or for locally advanced disease)
* No other concurrent chemotherapy
* Prior radiofrequency ablation allowed provided the following are true:

  * At least 4 weeks since prior radiofrequency ablation
  * Evidence of new tumor growth since therapy
* No prior radiotherapy to 25% or more of the bone marrow
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* Prior embolization allowed provided the following are true:

  * At least 4 weeks since prior embolization
  * Evidence of new tumor growth since therapy
* No prior pemetrexed disodium
* No aspirin or nonsteroidal anti-inflammatory drugs for at least 2 days (5 days for long-acting agents [e.g., piroxicam]) before, during, and for at least 2 days after administration of pemetrexed disodium
* No concurrent cyclo-oxygenase-2 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-01; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Survival after 6 months of treatment | Up to 6 months

SECONDARY OUTCOMES:
Response as assessed by RECIST criteria every 8-16 weeks | Up to 16 weeks
Toxicity as assessed by CTC v3 every 4 weeks | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (41):
- United States (41):
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Rutherford Hospital, Rutherfordton, North Carolina
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Alberts SR, Foster NR, McWilliams RR, et al.: NCCTG phase I/II trial (N9943) of gemcitabine and pemetrexed in patients with unresectable or metastatic biliary tract carcinoma and gallbladder carcinoma: interim results. [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-149, 2007.
- [Result] Alberts SR, Sande JR, Foster NR, Quevedo FJ, McWilliams RR, Kugler JW, Fitch TR, Jaslowski AJ. Pemetrexed and gemcitabine for biliary tract and gallbladder carcinomas: a North Central Cancer Treatment Group (NCCTG) phase I and II Trial, N9943. J Gastrointest Cancer. 2007;38(2-4):87-94. doi: 10.1007/s12029-008-9037-8. Epub 2008 Nov 21. PMID 19023677
- [Result] McWilliams RR, Foster NR, Quevedo FJ, et al.: NCCTG phase I/II trial (N9943) of gemcitabine and pemetrexed in patients with biliary tract or gallbladder carcinoma: phase II results. [Abstract] J Clin Oncol 25 (Suppl 18): A-4578, 2007.